CLINICAL TRIAL: NCT07396909
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single and Multiple Doses of MT-701 in Healthy Participants
Brief Title: A First-in-Human Single and Multiple Ascending Dose Study of MT-701
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mirador Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: MT-701-101
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers
Keywords: MT-701; Phase 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1- Single Ascending Dose (Experimental): To assess the safety and tolerability of single intravenous/subcutaneous dose of MT-701.
  Interventions: Drug: MT-701
- Part 2- Multiple Ascending Dose (Experimental): To assess the safety and tolerability of multiple intravenous/subcutaneous doses of MT-701.
  Interventions: Drug: MT-701

INTERVENTIONS:
Drug: MT-701 — MT-701

SUMMARY:
First-in-human study to evaluate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of single and multiple doses of MT-701 in healthy participants.

DETAILED DESCRIPTION:
This is a first-in-human study of MT-701, a biologic therapy. The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of single and multiple doses of MT-701 in healthy participants. The data obtained from this study will inform further development of MT-701.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (of non-childbearing potential only) participants between 19 and 55 years of age (inclusive) at the time of signing informed consent.
2. Female participants must be of nonchildbearing potential, defined as postmenopausal or surgically sterile and have official documentation, at least 6 months prior to the first dose.
3. Male participants must use highly effective forms of contraception during sexual intercourse with female partners of childbearing potential. A non-vasectomized, male subject must agree to use a condom with a chemical barrier method.
4. Good general health.
5. Able to provide written informed consent and understand and comply with the requirements of the study

Exclusion Criteria:

1. History or presence of any clinically significant organ system disease.
2. Abnormal laboratory assessments, physical exam of ECG outside the normal range that is judged by the Investigator to be clinically significant.
3. History of alcohol or drug abuse within the past 24 months.
4. Current use or history of regular tobacco or nicotine-containing products within 3 months prior to screening.
5. Administration of any prescription drug within 21 days of study drug administration; or over-the-counter drug within 7 days of study drug administration.
6. Administration or use of any investigational drug or device within 30 days preceding the first does of study drug administration.
7. Blood donation within 60 days prior to dosing or plasma donation within 14 days prior to dosing.
8. Sensitivity to any of the study drugs, or components thereof, or drug or other allergy that in the opinion of the Investigator or Sponsor Medical Monitor, contraindicates participation in the study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male and female (of non-childbearing potential only)
Enrollment: 78 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with non-SAEs and SAES | Up to 14 days post dose
  Incidence of adverse events, clinically significant laboratory abnormalities, clinically significant electrocardiogram, vital signs, and physical examination abnormalities.

CONTACTS AND LOCATIONS:
Locations (1):
- Mirador Clinical Department, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No